CLINICAL TRIAL: NCT05446337
Title: Diabetic Foot Care and Limb Preservation Pathway: Developmental Evaluation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-6156; PHSTE202201 (Other: Program for Health System and Technology Evaluation)
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Diabetic Foot; Lower Limb Wound; Diabetes; Amputation
Keywords: Developmental Evaluation; Care Pathway; Mixed-Methods Study
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients and Informal Care Givers: Individuals living with diabetes who are receiving or have received care through the Diabetes Foot Care and Limb Preservation Pathway at various stages of the care pathway including screening & prevention, wound care treatment, surgery and monitoring.
  Interventions: Other: Open-Ended Semi-Structured Interview
- Healthcare Providers: Medical, Nursing, and other allied healthcare providers including chiropodists, physiotherapists, occupational therapists, social workers, and nutritionists.
  Interventions: Other: Open-Ended Semi-Structured Interview
- Stakeholders: Individuals external and internal involved in clinical care, continuity of care, and policy-making including but not limited to senior hospital leadership, decision support, and researchers and policy decision-makers.
  Interventions: Other: Open-Ended Semi-Structured Interview

INTERVENTIONS:
Other: Open-Ended Semi-Structured Interview — Examine the participation and engagement in the Diabetic Foot Care and Limb Preservation Pathway design and implementation; identifying barriers and facilitators of the process

SUMMARY:
University Health Network (UHN), working together with local primary care practitioners, patients, and community healthcare services is developing a Diabetic Foot Care and Limb Preservation Care pathway. Our goal is to improve foot care for individuals living with diabetes. This study is using a method called developmental evaluation to help map out the system and to provide information in real-time so that the pathway can be adapted and respond to what is learned. The investigators are going to explore different factors (facilitators and barriers) and processes, which help or hinder the development, implementation, and adoption of the pathway. The investigators are also going to find out about the patient and provider's experiences with diabetic foot care, wound care, limb preservation, and amputation. Finally, the study team is going to look at value-based health care for the diabetic foot care pathways and document healthcare resource utilization, costs, and outcomes. The study team will conduct interviews of stakeholders, including patient representatives, and will examine the participation and engagement in the pathway, identifying barriers and facilitators of the process. Once the pathway has started, the study team will look at the way the care is delivered and satisfaction through surveys to patients and practitioners. The study team will also ask about patients' quality of life and their ability to manage diabetes. The study will aim to answer three key questions: What is happening? Why is it happening? and, What are reasonable prospects, and tools for change? The entire study is anticipated to take 3 years to complete.

DETAILED DESCRIPTION:
This study is a mixed-methods developmental evaluation study whose objectives are to:

1. Explore different factors (facilitators and barriers) and processes, which facilitate or impede the development, implementation, and adoption of Diabetes Foot Care and Limb Preservation Pathways using a multi-level framework.
2. Examine the patient and provider experiences with diabetic foot care, wound care, limb preservation, and amputation at UHN and the primary care settings and patient-level outcomes.

The developmental evaluation will consist of an initial component. Further quantitative and qualitative measures will be incorporated into the developmental evaluation as the Diabetic Foot Care and Limb Preservation Pathway develops.

1. Pathway Design & Implementation Case Study This qualitative research component will be completed through ethnographic fieldwork and the conduct of semi-structured interviews of stakeholders, including patient representatives, and will examine the participation and engagement in the Diabetic Foot Care and Limb Preservation Pathway design and implementation, identifying barriers and facilitators of the process. The study team will interview and observe three types of participants: patients and informal caregivers; healthcare providers including program service providers; stakeholders including hospital leadership and policy decision-makers. The research team will also attend meetings and collect and review documents and materials circulated as a part of the pathway development. In addition, social network analysis (SNA) may also be conducted as a part of this component to examine the interaction between stakeholders as well as the organizational dynamics and the fidelity of the intervention.

This study will be conducted in both the community and hospital settings at the University Health Network at Toronto General Hospital, Toronto Western Hospital, The Michener Institute of Education, Toronto Western Hospital Family Health Team (FHT) South Riverdale Community Health Centre, Primary Care Practices participating in the Seamless Care for Optimizing Patient Experience (SCOPE) and will be supported Nurse Navigators and by an Integrated Comprehensive Care (ICC) and associated homecare services.

ELIGIBILITY:
Inclusion Criteria:

Patients and Informal Caregivers:

* Diabetes (Type 1 and Type 2) receiving care within the Diabetes Foot Care and Limb Preservation Pathway
* Outpatient or inpatient care setting

Non-Patient Participants:

* Healthcare providers providing care
* Stakeholders supporting the clinical pathway development through University Health Network.
* In the early phases of the project a broader audience who may not be involved in the explicit design, outside of those that are designing the program, and may include external and internal stakeholders involved in clinical care, continuity of care, policy decision-making, patients, and caregivers.

Exclusion Criteria:

- Not able to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals from the Greater Toronto Area (GTA) that are involved with the Diabetes Foot Care and Limb Preservation Pathway through UHN either as patients and their caregivers, healthcare providers, or stakeholders.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Facilitators and Barriers | 9 months
  Key factors related to system readiness and implementation of the Diabetes Foot Care and Limb Preservation pathway

SECONDARY OUTCOMES:
Experience with Care | Duration of evaluation
  Experiences with diabetic foot care, wound care, limb preservation and amputation at UHN and the primary care settings and patient-level outcomes
Value-Based Healthcare | Duration of evaluation
  Potential of implementing value-based health care diabetic foot care pathways and document healthcare resource utilization, costs and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Valeria E. Rac, MD, PhD, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No